CLINICAL TRIAL: NCT02892929
Title: Effect of Motivational Interview as a Strategy in the Reduction of Blood Pressure in Hypertensive Patients in Specialist Clinic- Randomized Clinical Trial.
Brief Title: Effect of Motivational Interview as a Strategy in the Reduction of Blood Pressure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-0225
Record Dates: First submitted 2016-08-24; First posted 2016-09-08 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Hypertension
Keywords: Motivational Interviewing; Hypertension; Nursing; Randomized Controlled Trial; Life Style
MeSH Terms: conditions — Hypertension | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interviewing (Experimental): The motivational interview is a style of care that evokes the patient their motivations to make behavioral changes in the interests of their own health. It is a technique centered in patient to explore and resolve their ambivalence to modify unhealthy behavior.
  Interventions: Behavioral: Motivational interviewing
- Prescriptive Consultation (Active Comparator): Prescriptive consultation is the Methodology usual consultation. In this type of consultation the health professional who plans the action plan for the patient and determines how it will be the patient's lifestyle modification.
  Interventions: Behavioral: Prescriptive Consultation

INTERVENTIONS:
Behavioral: Motivational interviewing — The approach combines the principles of patient-centered care with strategies to motivate the change.
  Since the first appointment, Motivational Interviewing techniques will be used aiming to work the ambivalence that is to seek treatment and modify the unhealthy behavior. From the second encounter until the appointment of 120 days, the participants will be subjected to individual encounters in which the MI approach will be applied focusing on behavior change.
  Arms: Motivational Interviewing
Behavioral: Prescriptive Consultation — Prescriptive consultation is the Methodology usual consultation, in which the patient has little room to express themselves and the health professional who determines what and how the patient will hold the care of your health.
  Arms: Prescriptive Consultation

SUMMARY:
This randomized clinical trial was designed to test the effectiveness of Motivational Interviewing in lowering blood pressure during six months follow-up.

DETAILED DESCRIPTION:
The lead researcher is a cardiovascular nurse specialist with 10 years of experience in the care of patients with heart disease and she will be responsible for the application of the Motivational Interviewing (MI) technique in the appointments for the intervention group. She also participated in an intensive workshop about MI, which followed the recommendations of the Motivational Interviewing Network of Trainers19 in 2013, and more recently, in 2015 and 2016, she participated in two workshops on advanced MI techniques. During the study there will be monthly supervision with another specialist. The training and the supervision will be the responsibility of a PhD researcher in Psychiatry with consistent experience on Motivational Interviewing and training conducted in the United States with Miller and Rollnick.

The sample size was calculated with WinPepi 11.20 software. Sample size was estimated in 100 patients, 50 in the intervention group (IG) and 50 in the control group (CG), considering a difference of 8 mmHg between groups, standard deviation of 14 mmHg, 80% power, and alpha of 0.05. Adding 20% of losses the sample will have 120 patients, 60 for each group.

Hypertension outpatients of Hospital de Clínicas de Porto Alegre (HCPA) will be identified by the appointment book and invited to participate in the study through telephone calls. The first appointment will consist in obtaining the ICF and confirmation of eligibility. After ICF's signing and confirmation of eligibility, the patient will be randomized to one of the groups. Participants of both groups will attend monthly appointments: first appointment (D0), appointment of 30, 60, 90, 120, and 150 days, totaling six individual encounters, previously arranged in the Clinical Research Center (CRC) of HCPA, with an average duration of 30 minutes.

The randomization list was generated through the website www.randomization.com. The list will be in possession of a professional of the research group, however non-participant of this project. The allocation group of each patient will be hidden by opaque envelopes of identical appearance.

The researcher responsible for the application of the MI technique and the one responsible for the conduct of conventional appointments will be blinded to the outcomes of the study; therefore, the application of structured questionnaires, scales, and assessment of other variables of the study will be carried out by a researcher unblinded to the outcomes.

Statistical analysis:

Continuous variables will be expressed as mean standard deviation or median and interquartile range (25 and 75 percentile). Categorical variables will be expressed in absolute and percentage numbers. Chi-square will be used for associations between sociodemographic and clinical variables with the scores of the Self-Care Scale. The comparison of the quantitative variables between groups will be conducted by the Student's t-test or Mann-Whitney test, according to data's distribution. The values of systolic blood pressure (SBP) and diastolic blood pressure (DBP) during the study, as well as the scores of the Self-Care Scale will be analyzed by the Generalized Estimating Equations (GEE) with Bonferroni correction. The pressure differences between both groups during the treatment will be analyzed by ANOVA test for repeated measurements. Analysis of Covariance will be conducted to adjust possible differences regarding the basal pressure. The 5% level of significance will be adopted and the data will be analyzed in the Statistical Package for the Social Sciences (SPSS) v.20 (Chicago, Illinois, USA).

ELIGIBILITY:
Inclusion Criteria:

* Regular monitored in the hypertension outpatient clinic of HCPA for more than six months

Exclusion Criteria:

* Evident change in cognitive function, such as intellectual disability and dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
The reduction of at least 8 mmHg in systolic blood pressure and changes in diastolic blood pressure and mean blood pressure. | 6 months
  Measured by ABPM-24 h in the first and last protocol appointments

SECONDARY OUTCOMES:
regular use of antihypertensive medications. (Medication assessment questionnaire-MAQ) | 6 months
  The study also included the Medication Assessment Questionnaire (MAQ), is a four-item self-report adherence scale developed by Morisky, Green, and Levine to assess medication adherence. This scale is based on the understanding that lack of adherence to drug therapy could occur in one or all of several ways: forgetting, carelessness, discontinuation of medication when feeling better, or initiation of drug use when feeling worse. This scale is scored from 0 to 4, with lower scores reflecting higher adherence.
improvement of adherence to a low-sodium diet. (Dietary Sodium Restriction Questionnaire - DSRQ) | 6 months
  Scale that measures the adherence to a low-sodium diet.
adherence to self-care behaviors. (Self-care of hypertension Inventory SC-HI) | 6 months
  The self-care evaluation was performed using the Self-care of hypertension Inventory (SC-HI), which has proven validity and reliability for this purpose in hypertensive patients. This scale, based on the Middle Range Theory of Self-Care in Chronic Illness, was developed for a group of U.S. investigators and has since been translated and adapted for use in Brazil. The SC-HI measures three dimensions: self-care maintenance, consisting of those behaviors aimed at maintaining and monitoring disease stability; self-care management, i.e., the patient's response to the signs and symptoms of hypertension; and self-care confidence, i.e., self-efficacy in managing the two other domains. The SC-HI has a standardized score between 0-100. Higher score meaning better self-care.
Increase or maintenance of physical activity (International Physical Activity Questionnaire - IPAQ) | 6 months
  Questionnaire that mesures the physical activity.
weight reduction | 6 months
  Was measured at the baseline and final evaluation.
evaluation of changes in daytime sleepiness. (Epworth Sleepiness Scale) | 6 months
  Scale that measures the changes in daytime sleepiness.
Cessation smoking. (Questionnaire with questions about the amount of cigarettes smoked per week ) | 6 months
  That will be asked for the patients about the cessation smoking at baseline and at the final evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Graziella B Aliti, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silveira LCJ, Aliti GB, Da Silva EM, Pimentel RP, Gus M, Rabelo-Silva ER. Effect of motivational interviewing in hypertensive patients (MIdNIgHT): study protocol for a randomized controlled trial. Trials. 2019 Jul 9;20(1):414. doi: 10.1186/s13063-019-3486-1. PMID 31288854